CLINICAL TRIAL: NCT04818320
Title: Efficacy of Favipiravir in High Risk COVID-19 Patients: A Randomised, Open-label, Multicenter Clinical Trial
Brief Title: Favipiravir in High-risk COVID-19 Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Penang Hospital, Malaysia (Other Government)
Collaborators: Enche' Besar Hajjah Khalsom Hospital (Unknown); Jasin Hospital (Unknown); Kepala Batas Hospital (Other Government); Melaka Hospital (Unknown); Permai Hospital (Unknown); The Queen Elizabeth Hospital (Other); Raja Perempuan Zainab II Hospital (Unknown); Raja Permaisuri Bainun Hospital (Unknown); Sultanah Aminah Hospital (Unknown); Hospital Sultanah Nur Zahirah, Kuala Terengganu (Other Government); Sungai Buloh Hospital (Unknown); Tampin Hospital (Unknown); Tengku Ampuan Afzan Hospital (Unknown); Tuanku Fauziah Hospital (Unknown); Tuanku Jaafar Hospital (Unknown); Tumpat Hospital (Unknown); Institute for Clinical Research (Other); Tawau Hospital (Unknown); Hulu Terrengganu Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Favirpiravir-A1
Record Dates: First submitted 2021-03-24; First posted 2021-03-26 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — favipiravir

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Favipiravir (Experimental): Favipiravir treatment group (with standard of care),
  Interventions: Drug: Favipiravir
- Control (No Intervention): No favipiravir given. Standard of care only

INTERVENTIONS:
Drug: Favipiravir — Day 1: 1800mg BD, day 2-5: 800mg BD
  Arms: Favipiravir

SUMMARY:
The study aims to investigate the efficacy of favipiravir in high-risk COVID-19 patients. The study population includes symptomatic mild-to-moderate COVID-19 inpatients, within first 7 days of illness, who are 50 years old and above, and have 1 or more comorbidities. The study is designed as a randomised, open-label, multicenter clinical trial where the patients are randomised 1:1 to groups receiving favipiravir (5 days) versus no favipiravir.

ELIGIBILITY:
Inclusion Criteria:

* Patients are eligible to be included in the study only if they fulfil ALL the following criteria:
* RT-PCR confirmed COVID-19 cases
* Aged 50 years and above, AND have one or more co-morbidities
* Within the first 7 days of illness (from symptom onset)
* Mild to moderate clinical severity

Exclusion Criteria:

* Asymptomatic stage 1 patients
* Patients with SpO2 less than 95% without oxygen therapy
* Patients who needs oxygen supplements
* Patients with concomitant bacterial or fungal infection (confirmed by culture) prior to initiation of study
* Patients with congestive heart failure
* Patients with severe hepatic impairment (>Grade 3: ALT >10 times of upper normal limit)
* Impaired kidney function (creatinine clearance according to Cockcroft-Gault formula less than 30 ml/min) at the time of screening.
* Malabsorption syndrome or other clinically significant gastrointestinal disease that may affect absorption of the study drug (non-correctable vomiting, diarrhea, ulcerative colitis, and others).
* Pregnant or nursing women or women planning pregnancy.
* Female patients who cannot consent to contraceptive use of oral contraceptives, mechanical contraceptives such as intrauterine devices or barrier devices (pessaries, condoms), or a combination of these devices from the start of favipiravir administration to 7 days after the end of favipiravir administration
* Male patients whose partner cannot agree to use the contraception method described in (9)
* Patients with a history of gout or on treatment for gout or hyperuricemia
* Patients receiving immunosuppressants
* Patients who received interferon or drugs with reported antiviral activity against COVID-19 (hydroxychloroquine sulfate, chloroquine phosphate, lopinavir-ritonavir combination) within 7 days of illness.
* Patients in whom this episode of infection is a recurrence or reinfection of COVID-19 infection
* Patients who have previously received favipiravir
* Patients who are not able to provide written consent by themselves
* Other patients judged ineligible by the principal investigator or sub-investigator

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2021-02-16 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-13 (Actual)

PRIMARY OUTCOMES:
Need for oxygen supplement | Day of discharge/day 28 of treatment (if still hospitalized)
  Drop in SPO2 in room air to <95% or requiring supplemental oxygen to maintain SPO2≥95%

SECONDARY OUTCOMES:
Difference in the number of patients admitted to ICU | Day of discharge/day 28 of treatment (if still hospitalized)
Difference in the number of patients requiring mechanical ventilation | Day of discharge/day 28 of treatment (if still hospitalized)
Changes in the length of ICU stay | Day of discharge/day 28 of treatment (if still hospitalized)
Changes in in-hospital mortality rate | Day of discharge/day 28 of treatment (if still hospitalized)

CONTACTS AND LOCATIONS:
Locations (1):
- Penang General Hospital, George Town, Pulau Pinang, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chuah CH, Chow TS, Hor CP, Cheng JT, Ker HB, Lee HG, Lee KS, Nordin N, Ng TK, Zaid M, Zaidan NZ, Abdul Wahab S, Adnan NA, Nordin N, Tee TY, Ong SM, Chidambaram SK, Mustafa M; Malaysian Favipiravir Study Group. Efficacy of Early Treatment With Favipiravir on Disease Progression Among High-Risk Patients With Coronavirus Disease 2019 (COVID-19): A Randomized, Open-Label Clinical Trial. Clin Infect Dis. 2022 Aug 24;75(1):e432-e439. doi: 10.1093/cid/ciab962. PMID 34849615